CLINICAL TRIAL: NCT00423345
Title: Colon Investigation With Barium Enema, CT Colonography and Colonoscopy: A Prospective Registration of Indications, Delay and Procedure Results.
Brief Title: Colon Investigation - Factors Determining Choice of Procedure
Status: Terminated | Type: Observational
Why Stopped: One of the examinations (double contrast baium enema) became outdated in Norway
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Geir Hoff, Physician, head of gastroenterology, Notodden Hospital, Sykehuset Telemark
Other Study IDs: 23504
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Irritable Colon; Colorectal Cancer; Inflammatory Bowel Disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Registration of patients referred for colon investigation by barium enema, CT colonography and colonoscopy in two hospitals and one radiology centre in Telemark, Norway, for a period of minimum six months. Indications, delay and results of procedure will be recorded.Hypothesis: Choice of procedure for colon investigation is not based solely on clinical indication, but factors like delay, patient preference, lack of knowledge about the the procedures by the referring physician may have a decisive influence. The study will also analyse the correlation between patients symptoms, clinical findings and laboratory results and major pathology findings by colon investigation. Further, delay from patient´s first symptoms to finally diagnosis by colon investigation will also be registered and analysed.

DETAILED DESCRIPTION:
see extensive protocol in Norwegian

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to colon investigation
* Patients must be 18 years or older

Exclusion Criteria:

* Patients not able to give a written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for colonoscopy, barium enema or CT Colonoscopy and willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2006-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
findings compared across investigation modes | events by dec 2014
  Findings by one investigation compared to other

SECONDARY OUTCOMES:
Delayed diagnosis of CRC | events by dec 2014
  Waiting times depending on accessibility of diagnostic methods

CONTACTS AND LOCATIONS:
Overall Officials: Stein Dahler, MD, Principal Investigator — Blefjell Hospital Notodden, Norway; Gert Huppertz-Hauss, MD, Principal Investigator — Telemark Hospital, Norway; Arne R Hovland, MD, Principal Investigator — Telemark Radiology center, Porsgrunn, Norway
Locations (3):
- Norway (3):
  - Telemark Radiology center, Porsgrunn, Telemark
  - Department of gastroentology, Telemark Hospital, Skien, Telemark
  - Department of gastroentology, Blefjell Hospital Notodden, Notodden

IPD SHARING:
Plan to Share IPD: No